CLINICAL TRIAL: NCT03447457
Title: Early Initiation of High-flow Nasal Cannula Oxygen Therapy in Patients With Acute Respiratory Failure in the Emergency Department: A Before-after Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Collaborators: Centre Hospitalier de Niort (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: FLORAL-ER
Record Dates: First submitted 2018-02-19; First posted 2018-02-27 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Acute Respiratory Failure

STUDY DESIGN:
Intervention Model Description: FLORAL-ER is a before/after study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard oxygen group (Other): Patients are treated with standard oxygen delivered through nasal cannula, face mask or non-rebreathing reservoir
  Interventions: Device: Standard oxygen
- High-flow oxygen group (Other): Patients are treated with high-flow nasal cannula oxygen continuously applied via large-bore nasal prongs with a gas flow rate of 50 L/min
  Interventions: Device: High-flow oxygen

INTERVENTIONS:
Device: High-flow oxygen — HFNC is continuously applied via large-bore nasal prongs with a gas flow rate of 50 L/min and a FiO2 adjusted to maintain a pulse oxymetry at least 92%
  Other Names: High-flow nasal cannula oxygen therapy
  Arms: High-flow oxygen group
Device: Standard oxygen — nasal cannula, face mask or non-rebreathing reservoir mask
  Arms: standard oxygen group

SUMMARY:
The aim of the study is to compare the efficiency on respiratory failure regression of high-flow nasal oxygen therapy versus standard oxygen in patients admitted to the ED for de novo acute respiratory failure.

DETAILED DESCRIPTION:
Prospective observational before-after study at the ED in two French centers.

Selection of patients with acute hypoxemic respiratory failure at the ED.

Application of oxygen strategy according to the period:

* before period: standard oxygen delivered through nasal cannula, face mask or non-rebreathing reservoir mask, with a flow rate adjusted to maintain a pulse oxymetry of at least 92%.
* after period: high-flow oxygen therapy continuously applied via large-bore nasal prongs with a gas flow rate of 50 L/min and a FiO2 adjusted to maintain a pulse oxymetry at least 92%.

ELIGIBILITY:
Inclusion Criteria:

* de novo acute respiratory failure cowith the following criteria: a respiratory rate > 25 b/min, or signs of increased work of breathing.

Main exclusion Criteria:

* cardiogenic pulmonary edema,
* acute exacerbation of chronic lung disease, respiratory acidosis (pH < 7.35 and PaCO2 > 50 mm Hg),
* hemodynamic instability
* Glasgow Coma Scale score of 12 points or less,
* an urgent need for endotracheal intubation,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
complete regression of respiratory failure | one hour after initiation of oxygen strategies
  respiratory rate less than 25 breaths per minute and regression of signs of increased work of breathing

CONTACTS AND LOCATIONS:
Overall Officials: Jean MACE, MD, Study Director — Centre Hospitalier de Niort
Locations (2):
- France (2):
  - CHG de Niort, Niort
  - CHU Poitiers, Poitiers

IPD SHARING:
Plan to Share IPD: No